CLINICAL TRIAL: NCT01393249
Title: PEG-Asparaginase Associated Pancreatitis, Hepatotoxicity and Hyperlipidemia in Children With ALL
Acronym: AAP2008
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Kjeld Schmiegelow, Professor, Rigshospitalet, Denmark
Other Study IDs: RR240778PEGASP; H2-2010-002 (Registry Identifier: VEK RegionH)
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Acute Lymphoblastic Leukemia; Pancreatitis
Keywords: Acute Lymphoblastic Leukemia; Pediatric; Asparaginase; Pancreatitis
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALL, Asparaginase, pancreatitis: Patients that have been scanned and have had blood tests

SUMMARY:
The purpose of this study is to create a model enabling us to predict pancreatitis, hyperlipidemia and hepatotoxicity during treatment with PEG-Asparaginase in children with Acute Lymphoblastic Leukemia.

DETAILED DESCRIPTION:
Leukemia is the leading cause of cancer in children in Europe and the U.S. with an annual incidence of appoximately 3,5 cases per 100.000 children 0-14,9 years.

Although the rate of cure has increased significantly, treatment is still unsuccesfull in appoximately 20 % of the patients. There is great variation in the how the individual patient processes the different chemotherapeutic agents. Furthermore there is a signifikant difference regarding the severity of sideeffects and toxicities. So far it has not been possible to predict which patients are at speciel risk of developing toxicities.

Acute pancreatitis is a severe sideffect/toxicity when treating ALL. Patients are at risk of developing pancreatitis, because of the drug Asparaginase. The condition can not be prevented and in severe cases, e.g. hemorhaggic pancreatitis the only solution is to discontinue the drug, in spite of the fact that Asparaginase is on of the most important drugs when treating leukemia.

In the current study we will map the occurence of pancreatitis, hepatotoxicity and hyperlipidemia among approximately 1000 children and adolescents with leukemia. This study is unique because it is the largest study of its kind regarding Asparaginase associated pancreatitis. Among other things it will involve extensive genetic analysis.

We believe that this study will improve the possibilities, not only, for individualized treatmentVi mener at dette studie vil forbedre mulighederne for individ orienteret behandling, but also for other studies like this regarding other toxicities in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* IR- or SR- type ALL, and treatment with Peg-Asparaginase

Exclusion Criteria:

* HR ALL, and changing subgroup from IR or SR to HR

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 1-17.9, diagnosed with ALL and undergoing treatment with Peg-Asparaginase.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Risk of pancreatitis | During asparaginase therapy
  Risk of pancreatitis in relation to host genomic variants, inflammatory markers and ultrasound changes in the weeks prior to clinical pancreatitia

SECONDARY OUTCOMES:
Course of pancreatitis | In the months following pancreatitis
  Risk of complications, specifically cysts, pain and diabetes in the months following pancratitis.
  Risk of 2nd episode of pancreatitis if reexposed to asparaginase

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Schmiegelow, M.D., Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark